CLINICAL TRIAL: NCT06736444
Title: Efficacy of Brief Interventions to Reduce Comorbid Alcohol and Cannabis Misuse and Sleep Impairment in Young Adults (Rest-Up RCT)
Brief Title: Brief Interventions to Reduce Comorbid Alcohol and Cannabis Misuse and Sleep Impairment in Young Adults (Rest-Up RCT)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Mary Larimer, Professor, Department of Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00019900; 1R01AA031409-01A1 (NIH)
Record Dates: First submitted 2024-12-13; First posted 2024-12-16 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Insomnia; Alcohol Use; Marijuana Use
Keywords: Insomnia; Alcohol Use; Marijuana Use; Young Adults
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Alcohol Drinking; Marijuana Use | interventions — Ethanol; Mass Screening; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BASICSSLEEP (Experimental): The BASICSSLEEP intervention will integrate BASICS feedback and the Motivational Interviewing (MI) process described in the BASICS arm with Brief Behavioral Therapy for Insomnia (BBTI) content and materials. The BASICS + SLEEP intervention will be implemented in 2 sessions of 45-75 minutes and 2 telephone booster sessions. The investigators will follow BBTI procedures, including provision of a physiological rationale for insomnia and the importance of behavioral strategies to regulate sleep; introduction of sleep hygiene; discussion of factors that can impede duration and quality of sleep; introduction of sleep restriction and stimulus control strategies and negotiation of an initial sleep restriction schedule; and follow-up evaluation of success and continued refinement to achieve sleep efficiency goals. Booster contacts serve as opportunities to adjust the sleep restriction schedule, problem-solve challenges, and further build motivation.
  Interventions: Behavioral: Brief Behavioral Therapy for Insomnia (BBTI); Behavioral: Brief Alcohol Screening and Intervention for College Students (BASICS)
- BASICS+ (Active Comparator): The BASICS+ condition will meet for 2 sessions of 45-75 minutes. Content depends on the degree to which participants discuss the feedback, have questions, and/or explore behavior change options. Therapists review feedback components with participants, eliciting personally relevant reasons to change as domains are explored. When the participant is ambivalent about change, therapists work with them to explore and resolve that ambivalence. The method is non-confrontational and utilizes exploration of personalized graphic feedback (i.e., frequency, quantity, and peak use alongside perceived and actual norms for alcohol/MJ use) to increase motivation for change by highlighting ways alcohol and/or marijuana use could be incongruent with goals or values. Beliefs, expectations, and motives for use are discussed as are strategies to minimize risks and consequences. Booster sessions address questions and problem-solve challenges that have arisen since the session.
  Interventions: Behavioral: Brief Alcohol Screening and Intervention for College Students (BASICS)
- SLEEP (Active Comparator): The SLEEP intervention will be implemented in 2 sessions of 45-75 minutes and 2 telephone booster sessions. The investigators will follow BBTI procedures, including provision of a physiological rationale for insomnia and the importance of behavioral strategies to regulate sleep; introduction of sleep hygiene; discussion of factors that can impede duration and quality of sleep; introduction of sleep restriction and stimulus control strategies and negotiation of an initial sleep restriction schedule; and follow-up evaluation of success and continued refinement to achieve sleep efficiency goals.
  Interventions: Behavioral: Brief Behavioral Therapy for Insomnia (BBTI)
- Attention Control (Other): Attention Control (AC) participants complete all assessments (survey, daily, Fitbit, BAC) yoked to participants in the 3 active interventions, and attend the Zoom training to verify identity, orient to the Fitbit & BAC monitoring, and provide rationale and instructions for daily diaries. To better control for time and attention, AC participants attend 4 weekly Zoom check-ins (~20 minutes) in which clinically trained staff inquire about challenges encountered in monitoring, observations from monitoring, check in on mood/functioning, and provide referrals as needed. All conditions including AC receive community referrals to address substance uses, sleep, and mental health concerns. No participant is deprived of services; service use is tracked to assist with interpreting outcomes. AC participants will be offered BASICSSLEEP after completing 18-month follow-up.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Brief Behavioral Therapy for Insomnia (BBTI) — Brief Behavioral Therapy for Insomnia (BBTI) focuses primarily on stimulus control and sleep restriction as well as sleep hygiene recommendations delivered over 2 in-person sessions and 2 brief telephone boosters and is designed to be implemented by nonspecialists in primary care or other non-clinical settings. The intervention is manualized, and clients utilize sleep diaries and workbook assignments to consolidate recommendations.
  Arms: BASICSSLEEP; SLEEP
Behavioral: Brief Alcohol Screening and Intervention for College Students (BASICS) — Brief Alcohol Screening and Intervention for College Students (BASICS) is a manualized brief intervention targeting alcohol use and consequences among high risk drinkers and includes both personalized feedback regarding drinking norms, consequences, and motives for drinking, as well as protective behavioral skills for reducing heavy episodic drinking and related consequences. BASICS is delivered in a motivational interviewing (MI) style (Miller & Rollnick, 2002) to enhance intrinsic motivation to change drinking and implement protective behavioral strategies. BASICS has been adapted to target marijuana use and has been adapted for use with a variety of populations.
  Arms: BASICS+; BASICSSLEEP
Behavioral: Attention Control — Attention Control is comprised of 4 weekly 20-minute check-ins with a study therapists regarding the daily monitoring and mood/functioning. Referrals for additional services will be provided as needed.
  Arms: Attention Control

SUMMARY:
This study is designed to evaluate an integrated intervention to reduce alcohol and marijuana use and consequences and improve sleep among young adults with comorbid heavy episodic drinking, marijuana use, and sleep impairment.

DETAILED DESCRIPTION:
This study is designed to evaluate an integrated brief intervention to reduce alcohol and cannabis use and consequences and improve sleep among young adults (YA) with comorbid heavy episodic drinking (HED), cannabis misuse, and sleep impairment. HED in YA is an important public health problem; consequences include accidental injury and death, academic/work problems, unsafe and unwanted sex, and development of alcohol use disorders. Many YA with HED also use cannabis and experience increased harm as a result. Sleep impairment is common and problematic among YA, identified as one of 5 leading barriers to academic success for students and an important risk factor for mental health problems and suicide in YA. More than 75% of YA report frequent daytime fatigue, 27% extreme distress related to sleep problems, and more than 1 in 4 are at high risk for insomnia. Alcohol use has been linked to insomnia in adolescent, YA, and older adult populations, with bidirectional causal links between alcohol use and impaired sleep. Comorbidity of HED and sleep impairment is associated with increased consequences of alcohol use and exacerbates risk of accidents (including automobile accidents), impaired decision-making, and work and academic difficulties. Similar bidirectional relations exist with cannabis use and sleep, and co-use of these substances may be particularly harmful for sleep. Despite these risks, alcohol and cannabis prevention programs rarely target sleep directly, and the majority of YA sleep interventions either focus on sleep hygiene broadly in the absence of specific strategies to improve sleep or reduce alcohol/cannabis use or have insufficient sample size and duration to truly evaluate impacts on sleep or related comorbid alcohol or cannabis use. Building on the investigators' successful R34 intervention development project, the current study addresses these gaps by evaluating efficacy of integrating a brief sleep intervention (BBTI) with an efficacious brief alcohol and cannabis intervention (BASICS/Cannabis BMI) to increase magnitude and duration of effects on sleep and alcohol and cannabis misuse among a diverse community sample of YA with comorbid insomnia, HED, and cannabis use. Given bidirectional influences between sleep impairment and alcohol/cannabis misuse leading to significant public health challenges for this population, an efficacious integrated treatment is imperative. Impact will be evaluated in a RCT comparing efficacy of telehealth-delivered, integrated BASICSSLEEP to BASICS/BMI only (BASICS+), BBTI only (SLEEP), and Attention control (AC). Surveys and daily diaries will assess alcohol, cannabis, and sleep at baseline, post-treatment, 3-, 6-, 12-, and 18-months. Specific aims are: (1) Evaluate comparative efficacy of BASICSSLEEP, BASICS+, and SLEEP in reducing alcohol/cannabis use and consequences and improving sleep; (2) Evaluate moderators of efficacy for integrated and monotherapies; and (3) Use diary data to evaluate temporal sequencing of effects and duration/decay over time. Findings will remedy important gaps in the literature and result in a scalable, accessible new resource to address this important and costly comorbidity.

ELIGIBILITY:
Inclusion Criteria:

* Participants must: 1) be 18-24 years old; 2) reside in Washington State; 3) have valid email address; 4) score on the Insomnia Severity Index (ISI) of 10 or higher, indicating at least a moderate score (score of 2 or more) on one or more of the first three items of the ISI measuring difficulty falling asleep, staying asleep, or waking up too early; 5) report at least two heavy drinking episodes (4+ drinks for women /gender diverse, 5+ for men in a 2-hour period) in the past month; 6) have used cannabis 6+ times in the past month; and 7) did not participate in the R34 pilot feasibility trial on which the current RCT is based.

Exclusion Criteria:

* Participants that don't meet inclusion criteria and/or failure to consent to further participation.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Baseline, Post-Intervention (7 weeks post-Baseline), 3 Month Follow-up (3 months post-Baseline), 6 Month Follow-up (6 months post-Baseline), 12 Month Follow-up (12 months post-Baseline), 18 Month Follow-up (18 months post-Baseline)
  The Insomnia Severity Index is a 7-item measure that assesses the severity of both nighttime and daytime aspects of insomnia. Response options utilized a 5-point Likert scale ranging from 0-4 where "0" reflected low symptom endorsement and "4" reflected high symptom endorsement. Responses across the 7 items are summed to create a Total Score. Total Scores range from 0 to 28. Total scores of 0-7=No clinically significant insomnia, 8-14=subthreshold insomnia, 15-21=clinical insomnia (moderate severity), and 22-28=clinical insomnia (severe).
Patient-Reported Outcomes Information System Short Form v1.0 Sleep-Related Impairment 8a (PROMIS SF8 v1.0 SRI) | Baseline, Post-Intervention (7 weeks post-Baseline), 3 Month Follow-up (3 months post-Baseline), 6 Month Follow-up (6 months post-Baseline), 12 Month Follow-up (12 months post-Baseline), 18 Month Follow-up (18 months post-Baseline)
  The Patient-Reported Outcomes Information System Short Form v1.0 Sleep Related Impairment 8a (8-items) assesses self-reported perceptions of impairment due to sleep problems. Response options range from 1=Not at all to 5=Very much and are summed to create a raw score (range 8-40). Raw scores are transformed to T-scores with a population mean of 50 and a standard deviation (SD) of 10, where higher scores indicate greater impairment due to sleep problems. For example, a T-score of 60 is one SD worse than average, whereas a T-score of 40 is one SD better than average.
Quantity/Frequency/Peak Alcohol Use Index (QFP) peak item | Baseline, Post-Intervention (7 weeks post-Baseline), 3 Month Follow-up (3 months post-Baseline), 6 Month Follow-up (6 months post-Baseline), 12 Month Follow-up (12 months post-Baseline), 18 Month Follow-up (18 months post-Baseline)
  The Quantity Frequency Peak Alcohol Use Index was used to assess the peak number of standard drinks consumed on their heaviest drinking occasion over the previous month.
Quantity/Frequency/Peak Alcohol Use Index (QFP) quantity item | Baseline, Post-Intervention (7 weeks post-Baseline), 3 Month Follow-up (3 months post-Baseline), 6 Month Follow-up (6 months post-Baseline), 12 Month Follow-up (12 months post-Baseline), 18 Month Follow-up (18 months post-Baseline)
  The Quantity Frequency Peak Alcohol Use Index was used to assess typical drinking quantity using the number of drinks consumed during a typical drinking occasion over the previous month.
Quantity/Frequency/Peak Alcohol Use Index (QFP) frequency item | Baseline, Post-Intervention (7 weeks post-Baseline), 3 Month Follow-up (3 months post-Baseline), 6 Month Follow-up (6 months post-Baseline), 12 Month Follow-up (12 months post-Baseline), 18 Month Follow-up (18 months post-Baseline)
  The Quantity Frequency Peak Alcohol Use Index was used to assess the frequency of drinking over a typical week over the previous month. Response options range from 0=I do not drink at all to 7=Every day.
Daily Drinking Questionnaire (DDQ) | Baseline, Post-Intervention (7 weeks post-Baseline), 3 Month Follow-up (3 months post-Baseline), 6 Month Follow-up (6 months post-Baseline), 12 Month Follow-up (12 months post-Baseline), 18 Month Follow-up (18 months post-Baseline)
  The Daily Drinking Questionnaire assesses the typical number of drinks consumed on each day of a typical week over the previous month. Responses were summed to create a total score of overall number of standard drinks consumed over a typical week.
Rutgers Alcohol Problems Index | Baseline, Post-Intervention (7 weeks post-Baseline), 3 Month Follow-up (3 months post-Baseline), 6 Month Follow-up (6 months post-Baseline), 12 Month Follow-up (12 months post-Baseline), 18 Month Follow-up (18 months post-Baseline)
  The Rutgers Alcohol Problem Index (23 items) assessed negative consequences related to drinking. Two items were added to assess driving after drinking 2 or more drinks and 4 or more drinks. Response options range from 0=Never to 4=More than 10 times. Responses were summed to create a total score of problems experienced in the previous 3 months. Possible scores ranged from 0 to 100.

SECONDARY OUTCOMES:
Daily Marijuana Questionnaire | Baseline, Post-Intervention (7 weeks post-Baseline), 3 Month Follow-up (3 months post-Baseline), 6 Month Follow-up (6 months post-Baseline), 12 Month Follow-up (12 months post-Baseline), 18 Month Follow-up (18 months post-Baseline)
  The Daily Marijuana Questionnaire was used to assess hours high from cannabis use on each day over a typical week in the past month. Items were summed to create a total score of overall number of hours spent high during a typical week.
Marijuana-Related Consequences | Baseline, Post-Intervention (7 weeks post-Baseline), 3 Month Follow-up (3 months post-Baseline), 6 Month Follow-up (6 months post-Baseline), 12 Month Follow-up (12 months post-Baseline), 18 Month Follow-up (18 months post-Baseline)
  Marijuana Consequences were assessed with a 29-item measure assessing consequences related to marijuana use. Response options range from 0=Never to 4=More than 10 times. Scores are summed to create a total score of problems experienced in the previous 3 months. Possible scores ranged from 0 to 116.

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Larimer, Ph.D., Principal Investigator — University of Washington